CLINICAL TRIAL: NCT01255709
Title: CLINICAL STUDY-B3 FOR ASSESSMENT OF PHARMACOKINETICS, A Randomized, Evaluator-Blind, Single-Dose, Three Arm, Crossover,PK Study in Healthy Volunteers
Brief Title: Epinephrine Inhalation Aerosol USP, CLINICAL STUDY-B3 FOR ASSESSMENT OF PHARMACOKINETICS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: API-E004-CL-B3
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: Asthma; shortness of breath; wheezing
MeSH Terms: conditions — Asthma; Dyspnea; Respiratory Sounds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm T1 Primatene Mist HFA (Experimental): epinephrine inhalation aerosol, 90 mcg/inhalation, 12 inhalations over 6 minutes
  Interventions: Drug: Arm T1: Primatene Mist HFA
- Arm C Primatene Mist (Active Comparator): epinephrine inhalation aerosol, 220 mcg/inhalation, 12 inhalations over 6 minutes
  Interventions: Drug: Arm C: Primatene Mist (epinephrine inhalation aerosol, USP)
- Arm T2 Primatene Mist HFA (Experimental): epinephrine inhalation aerosol, 100 mcg/inhalation, 12 inhalations over 6 minutes
  Interventions: Drug: Arm T2: Primatene Mist HFA

INTERVENTIONS:
Drug: Arm T1: Primatene Mist HFA — epinephrine inhalation aerosol, 90 mcg/inhalation, 12 inhalations over 6 minutes
  Other Names: epinephrine inhalation aerosol
  Arms: Arm T1 Primatene Mist HFA
Drug: Arm T2: Primatene Mist HFA — epinephrine inhalation aerosol, 100 mcg/inhalation, 12 inhalations over 6 minutes
  Other Names: epinephrine inhalation aerosol
  Arms: Arm T2 Primatene Mist HFA
Drug: Arm C: Primatene Mist (epinephrine inhalation aerosol, USP) — epinephrine inhalation aerosol, 220 mcg/inhalation, 12 inhalations over 6 minutes
  Other Names: epinephrine inhalation aerosol
  Arms: Arm C Primatene Mist

SUMMARY:
This study examines the pharmacokinetic profile of Armstrong's proposed Epinephrine Inhalation Aerosol USP, an HFA134a propelled Metered Dose Inhaler (MDI) (E004), using a stable isotope deuterium-labeled epinephrine (epinephrine-d3) to differentiate the administered drug from the endogenous epinephrine, in healthy male and female adult volunteers.

DETAILED DESCRIPTION:
The current study is designed to complement and expand the previous PK studies, API-E004-CL-B and API-E004-CL-B2, with emphasis on lower E004 dose strengths (at 90 and 100 mcg per inhalation), for a more thorough evaluation of the E004 PK profiles. Safety of E004 will also be evaluated, under augmented dose conditions.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy at screening;
* Body weight ≥ 50 kg for men and ≥ 45 kg for women;
* Sitting blood pressure ≤ 135/90 mmHg;
* Demonstrating negative hIV, HBsAG and DCV-Ab screen tests;
* Women of child-bearing potential must be non-pregnant, non-lactating, and practicing a clinically acceptable form of birth control;
* Properly consented
* Other criteria apply

Exclusion Criteria:

* A smoking history of ≥10 pack-years, or having smoked within 6 months prior to Screening;
* Upper respiratory tract infections within 2 wk, or lower respiratory tract infection within 4 wk, prior to Screening;
* Any current or recent respiratory conditions that might significantly affect pharmacodynamic response to the study drugs;
* Known intolerance or hypersensitivity to the study MDI ingredients;
* Having been on other investigational drug/device studies, or donated blood, in the last 30 days prior to Screening;
* Other criteria apply

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics including maximum concentration and area under the curve | -30, 2, 5, 7.5, 10, 12.5, 15, 20, 25, 30, 45, 60, 90, 120, 240 and 360 min postdose.
  Samples will be analyzed with an established LC/MS/MS method, with a quantitative detection limit of 0.02 ng/mL, for both epinephrine-d3 and epinephrine-h3.
  * Mean Maximum concentration of epinephrine (Cmax for epinephrine)
  * Mean Area Under the Curve (AUC) for epinephrine
  * Time to maximum concentration (tmax) and Half life of the drug (t1/2)
  * Epinephrine concentrations versus time

SECONDARY OUTCOMES:
Vital Signs | within 30 min predose, at 30, 60 and 360 min postdose
  Systolic and Diastolic Blood pressure and heart rate
12-lead Electrocardiogram (ECG) | within 30 min pre-dose, and at 15 and 120 min post-dose
  12 lead ECG (Routine and QT/QTc intervals)
Telemetry ECG | within 30 min pre-dose, and during the initial 5 min post-dose
  Telemetry recording of heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Amphastar Pharmaceuticals, Inc.
Locations (1):
- Amphastar Study Site 1, Cypress, California, United States

REFERENCES:
- [Background] Pinnas JL, Schachtel BP, Chen TM, Roseberry HR, Thoden WR. Inhaled epinephrine and oral theophylline-ephedrine in the treatment of asthma. J Clin Pharmacol. 1991 Mar;31(3):243-7. doi: 10.1002/j.1552-4604.1991.tb04969.x. PMID 2019665
- [Background] Hendeles L, Marshik PL, Ahrens R, Kifle Y, Shuster J. Response to nonprescription epinephrine inhaler during nocturnal asthma. Ann Allergy Asthma Immunol. 2005 Dec;95(6):530-4. doi: 10.1016/S1081-1206(10)61014-9. PMID 16400891
- [Background] Warren JB, Doble N, Dalton N, Ewan PW. Systemic absorption of inhaled epinephrine. Clin Pharmacol Ther. 1986 Dec;40(6):673-8. doi: 10.1038/clpt.1986.243. PMID 3780129
- [Background] Cripps A, Riebe M, Schulze M, Woodhouse R. Pharmaceutical transition to non-CFC pressurized metered dose inhalers. Respir Med. 2000 Jun;94 Suppl B:S3-9. PMID 10919679
- [Background] Dickinson BD, Altman RD, Deitchman SD, Champion HC. Safety of over-the-counter inhalers for asthma: report of the council on scientific affairs. Chest. 2000 Aug;118(2):522-6. doi: 10.1378/chest.118.2.522. PMID 10936150
- [Background] Simons FE, Gu X, Johnston LM, Simons KJ. Can epinephrine inhalations be substituted for epinephrine injection in children at risk for systemic anaphylaxis? Pediatrics. 2000 Nov;106(5):1040-4. doi: 10.1542/peds.106.5.1040. PMID 11061773
- [Background] Kushner DJ, Baker A, Dunstall TG. Pharmacological uses and perspectives of heavy water and deuterated compounds. Can J Physiol Pharmacol. 1999 Feb;77(2):79-88. PMID 10535697
- [Background] Bondesson E, Friberg K, Soliman S, Lofdahl CG. Safety and efficacy of a high cumulative dose of salbutamol inhaled via Turbuhaler or via a pressurized metered-dose inhaler in patients with asthma. Respir Med. 1998 Feb;92(2):325-30. doi: 10.1016/s0954-6111(98)90116-0. PMID 9616533